CLINICAL TRIAL: NCT07210255
Title: A Randomized Controlled Multi-site Trial Evaluating SAINT for Postpartum Depression
Brief Title: SAINT in Postpartum Depression (PPD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Magnus Medical (Industry)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLN-0108; CDMRP-PR240070 (Other Grant/Funding Number: USAMRAA)
Record Dates: First submitted 2025-09-15; First posted 2025-10-07 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Postpartum Depression (PPD)
Keywords: SAINT; Stanford Accelerated Intelligent Neuromodulation Therapy; Repetitive Transcranial Magnetic Stimulation (rTMS); Intermittent Theta Burst Stimulation (iTBS); Noninvasive Brain Stimulation; Postpartum depression; Neuromodulation
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: This is a multisite, randomized controlled trial. This study has two phases, a blinded/acute phase in which participants are randomized to receive either 5 days of active or sham SAINT and a follow-up phase in which all participants will be followed for 6 months and may be eligible to receive 1 course of open-label active SAINT (5 days).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study monitors, SAINT treaters, research coordinators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active SAINT Stimulation (Active Comparator): Active SAINT stimulation will be applied to the left dorsolateral prefrontal cortex (L-DLPFC)
  Interventions: Device: SAINT Neuromodulation System
- Sham SAINT Stimulation (Sham Comparator): Sham (non-active) stimulation will be applied to the left dorsolateral prefrontal cortex (L-DLPFC).
  Interventions: Device: Sham SAINT Stimulation

INTERVENTIONS:
Device: SAINT Neuromodulation System — SAINT will be delivered via a MagPro X100 edition (MagVenture, Skovlunde, Denmark) TMS device equipped with a Cool-B65 A/P coil. The stimulation paradigm consists of 10 daily sessions (50 total sessions over 5 days) of SAINT stimulation (3-pulse 50-Hz bursts at 5-Hz for 2-second trains, with trains every 10 seconds), delivered with 50-minute inter-session intervals (10-minute sessions, 50-minutes in between sessions). Stimulation will be administered at 90% of the participant's resting motor threshold, with depth correction applied to adjust for the measured distance between the scalp and cortical surface. The stimulation target, the L-DLPFC, will be identified and localized by the study investigator using the Localite neuronavigation system.
  Other Names: SAINT NMS; SAINT
  Arms: Active SAINT Stimulation
Device: Sham SAINT Stimulation — Sham stimulation will be delivered using the MagVenture MagPro X100 TMS system with the Cool-B65 A/P coil and targeted to the L-DLPFC. The stimulation paradigm will be identical to the active SAINT stimulation with the exception that active stimulation will not be delivered.
  Arms: Sham SAINT Stimulation

SUMMARY:
This study is a large, multi-site clinical trial testing whether Stanford Accelerated Intelligent Neuromodulation Therapy (SAINT), a fast-acting form of repetitive transcranial magnetic stimulation (rTMS), can more effectively reduce symptoms of postpartum depression (PPD) compared to a sham treatment.

It will enroll 192 women within six months postpartum who are experiencing depression that has not improved with standard care, and will track their progress for up to six months. The trial's main goal is to see if SAINT leads to rapid improvement in depression, while also evaluating its safety, durability of benefit, and impact on mother-infant bonding.

DETAILED DESCRIPTION:
SAINT combines an accelerated rTMS stimulation protocol with individualized functional connectivity (FC)-based brain targeting. It has demonstrated dramatic remission rates of 80-90% in patients with treatment resistant depression (TRD) in 5 days or fewer of treatment. SAINT is FDA cleared for the treatment of major depressive disorder (MDD) in adult patients who have failed to achieve satisfactory improvement from prior antidepressant medication in the current episode.

This is a multi-site, randomized trial to assess SAINT versus sham stimulation for PPD in women who are non-responsive to standard of care treatment. This study will evaluate whether SAINT is superior to placebo in reducing symptoms of depression in PPD among women unresponsive to standard care. Unlike traditional treatments, SAINT is designed to provide rapid relief from depressive symptoms, potentially within just a few days. The rationale for this study is based on the need for a faster, more effective treatment option that can quickly stabilize the mental health of new mothers, allowing them to better care for their infants and themselves.

This study will primarily benefit women who have recently given birth and are struggling with a postpartum depression. These women often face intense emotional distress that can interfere with their ability to bond with their newborns and manage daily responsibilities. By offering a quicker route to recovery, SAINT has the potential to restore these mothers' mental health, enabling them to fully engage in their new role as parents. The study also aims to include a diverse population, ensuring that the benefits of SAINT are generalizable.

There are two phases in this study:

1. A blinded phase where participants will be randomized to receive 5 days of active SAINT, an accelerated and individualized form of rTMS, or a sham (placebo) treatment.
2. After the acute treatment, participants will enter the 6 month follow-up phase. During this phase, if participants experience worsening symptoms, they will be offered 1 course of active SAINT treatment. (5 days).

Total study duration for each participant is approximately 7.5 months.

ELIGIBILITY:
Inclusion Criteria:

1. Reproductive Women ages 18-45 at the time of consent.
2. Diagnosis of non-psychotic Major Depressive Episode (MDE) with peripartum onset as assessed through the Quick Structured Clinical Interview for DSM-5.
3. 0-12 months postpartum. Participants must be 0-12 months postpartum at screening and remain within 12 months postpartum at the 5-day post-treatment visit.
4. If currently taking an antidepressant medication and/or receiving psychotherapy must be on a stable regimen for 30 days at the time of enrollment.
5. Severe depression as measured by MADRS ≥20 at screening.
6. A good candidate for repetitive transcranial magnetic stimulation (rTMS) as determined by a physician.
7. Participants must be capable of giving informed consent. Participants must be proficient in English in order to comprehend study requirements.
8. Agree to use effective contraception in the postpartum period for the study duration.
9. Willing and able to comply with all study procedures, complete required assessments and visits, and be available for the duration of the study.

Exclusion Criteria:

1. Participant has attempted suicide in the last 6 months and/or expressed suicidal ideation with intent as determined by physician assessment at the time of enrollment.
2. Score of 6 on MADRS item 10 (high rating of suicidal ideation) at screening.
3. Participant has active psychosis per investigator assessment.
4. Participant with a primary lifetime diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder and/or obsessive-compulsive disorder.
5. Participant has an active eating disorder or substance use disorder in the past 6 months and/or has a positive urine toxicity screen that the Principal Investigator (PI) deems exclusionary.
6. Participant is using any exclusionary medications: high dose of benzodiazepines (>2mg lorazepam daily equivalent and/or >3 times per week) or medications that would interfere with treatment with TMS as per PI or designee discretion.
7. Participant has a history of untreated or insufficiently treated sleep apnea.
8. Participant has a history of significant neurologic disease, including developmental disability, dementia, Parkinson's or Huntington's disease, brain tumor, unexpected seizure/epilepsy disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma.
9. Any untreated major somatic illness such as hypertension/cardiovascular disease/diabetes/endocrine disorders etc.
10. Contraindications to receiving rTMS (e.g., metal in head, history of seizure, known brain lesion).
11. Contraindications to MRI (e.g., ferromagnetic metal in their body).
12. Currently pregnant.
13. History of receiving rTMS for any reason, as this may compromise blinding.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 192 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline and 5 days post-acute treatment
  The change in depression symptom severity will be measured by Montgomery-Åsberg Depression Rating Scale (MADRS), from baseline to 5 days post-treatment. Outcomes will be compared between the acute active SAINT and sham arms. Scores range from 0-60 (10 questions, each scored 0-6) with higher scores indicating a worsening of depressive symptoms and lower scores indicating better outcomes.

OTHER OUTCOMES:
Montgomery-Asberg Depression Rating Scale - Self Report (MADRS-S) | Baseline, 5 days post acute treatment through 6 months (180 days) post-treatment follow-up (assessed every 14 days).
  Durability of treatment will be assessed from immediately after treatment through six months (180 days) using the Montgomery-Åsberg Depression Rating Scale - Self Report (MADRS-S). The MADRS-S consists of 9 questions, each scored from 0 to 3, with a total score range of 0-27. Higher scores indicate greater depressive symptom severity, while lower scores indicate improvement in symptoms.
Treatment Adherence and Acceptability Scale (TAAS) | 5-day post acute treatment visit and if applicable, 5 days post open-label treatment visit.
  Treatment acceptance and adherence will be assessed using the 10-item Treatment Acceptance and Adherence Scale (TAAS). Each item is rated from 1 to 7, for a total score range of 10 to 70. Higher scores indicate greater treatment acceptance and adherence, while lower scores indicate poorer acceptance and adherence.
Mother-to-Infant Bonding Scale (MIBS) | Baseline, 1 month, 3 months, 6 months post-treatment
  An 8-item self-report questionnaire used to assess the early emotional bond between a mother and her infant. Each item is scored 0-3 with a score ranging from 0-24. Higher scores reflect greater bonding difficulties; lower scores reflect more positive bonding.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - UMass Chan Medical School, Worcester, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Medical University of South Carolina (MUSC), Charleston, South Carolina
  - University of Texas at Austin, Dell Medical School, Health Discovery Building, Austin, Texas

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality concerns. Aggregate study results will be made publicly available on ClinicalTrials.gov and through publications.

REFERENCES:
- [Background] Williams NR, Sudheimer KD, Bentzley BS, Pannu J, Stimpson KH, Duvio D, Cherian K, Hawkins J, Scherrer KH, Vyssoki B, DeSouza D, Raj KS, Keller J, Schatzberg AF. High-dose spaced theta-burst TMS as a rapid-acting antidepressant in highly refractory depression. Brain. 2018 Mar 1;141(3):e18. doi: 10.1093/brain/awx379. No abstract available. PMID 29415152
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538